CLINICAL TRIAL: NCT01468181
Title: A 52-Week, Open-Label, Long-Term Safety Study of LY2189265 in Combination With Monotherapy of Oral Antihyperglycemic Medications in Patients With Type 2 Diabetes Mellitus
Brief Title: A Study of LY2189265 in Japanese Participants With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13991; H9X-JE-GBDQ (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-11-07; First posted 2011-11-09 (Estimated); Results first posted 2014-12-16 (Estimated); Last update posted 2015-01-29 (Estimated); Status verified 2015-01

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes mellitus; Oral antihyperglycemic medications; Long-Term Safety; GLP 1; Glucagon like peptide 1
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dulaglutide; Sulfonylurea Compounds; Biguanides; Glycoside Hydrolase Inhibitors; 2,4-thiazolidinedione

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- LY2189265 + Sulfonylureas (SU) (Experimental): LY2189265: 0.75 milligrams (mg) administered subcutaneously (SC), once weekly for 52 weeks
  Participants were to continue on their stable, pre-study, physician-prescribed dose of SU monotherapy throughout the study.
  Interventions: Drug: LY2189265; Drug: Sulfonylureas (SU)
- LY2189265 + Biguanides (BG) (Experimental): LY2189265: 0.75 mg administered SC, once weekly for 52 weeks
  Participants were to continue on their stable, pre-study, physician-prescribed dose of BG monotherapy throughout the study.
  Interventions: Drug: LY2189265; Drug: Biguanides (BG)
- LY2189265 + alpha-glucosidase inhibitor (a-GI) (Experimental): LY2189265: 0.75 mg administered SC, once weekly for 52 weeks
  Participants were to continue on their stable, pre-study, physician-prescribed dose of a-GI monotherapy throughout the study.
  Interventions: Drug: LY2189265; Drug: alpha-glucosidase inhibitor (a-GI)
- LY2189265 + Thiazolidinedione (TZD) (Experimental): LY2189265: 0.75 mg administered SC, once weekly for 52 weeks
  Participants were to continue on their stable, pre-study, physician-prescribed dose of TZD monotherapy throughout the study.
  Interventions: Drug: LY2189265; Drug: Thiazolidinedione (TZD)
- LY2189265 + Glinides (Experimental): LY2189265: 0.75 mg administered SC, once weekly for 52 weeks
  Participants were to continue on their stable, pre-study, physician-prescribed dose of glinides monotherapy throughout the study.
  Interventions: Drug: LY2189265; Drug: Glinides

INTERVENTIONS:
Drug: LY2189265
  Other Names: Dulaglutide
Drug: Sulfonylureas (SU) — SU is a pre-study prescribed dose and is not being provided as part of the trial.
  Arms: LY2189265 + Sulfonylureas (SU)
Drug: Biguanides (BG) — Biguanides is a pre-study prescribed dose and is not being provided as part of the trial.
  Arms: LY2189265 + Biguanides (BG)
Drug: alpha-glucosidase inhibitor (a-GI) — a-GI is a pre-study prescribed dose and is not being provided as part of the trial.
  Arms: LY2189265 + alpha-glucosidase inhibitor (a-GI)
Drug: Thiazolidinedione (TZD) — TZD is a pre-study prescribed dose and is not being provided as part of the trial.
  Arms: LY2189265 + Thiazolidinedione (TZD)
Drug: Glinides — Glinides is a pre-study prescribed dose and is not being provided as part of the trial.
  Arms: LY2189265 + Glinides

SUMMARY:
This was a 52-week, multicenter, non-randomized, open-label, Phase 3 long-term safety study in participants with type 2 diabetes mellitus who have inadequate glycemic control with monotherapy of oral antihyperglycemic medication (OAM).

ELIGIBILITY:
Inclusion Criteria:

* Participants who have had a diagnosis of type 2 diabetes mellitus before screening
* Participants who have been taking SU (Glibenclamide, Gliclazide, Glimepiride), BG, TZD, a-GI or glinides monotherapy for at least 3 months before screening and have been on a stable dose for at least 8 weeks before screening
* Participants must have a qualifying HbA1c value of 7.0% to 11.0% at screening
* Participants who have a body mass index (BMI) of 18.5 to 35.0 kilograms per meter squared (kg/m^2)

Exclusion Criteria:

* Participants who have a diagnosis of type 1 diabetes
* Participants who have previously been treated with any other glucagon-like peptide-1 (GLP-1) analog within the 3 months before screening
* Participants who are currently taking insulin or have had previous insulin treatment within the 3 months before screening
* Participants who have obvious clinical signs or symptoms of pancreatitis, a history of chronic pancreatitis, or acute pancreatitis at screening, as determined by the investigator. Participants who have a serum amylase concentration ≥3 times the upper limit of the reference range and/or a serum lipase concentration ≥2 times the upper limit of the reference range, as determined by the central laboratory at screening
* Participants who have self or family history of medullary C-cell hyperplasia, focal hyperplasia, or medullary thyroid carcinoma (MTC)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 394 (Actual)
Dates: Start 2011-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM-5PM Eastern time (UTC/GMT - 5, hours, EST), Study Director — Eli Lilly and Company
Locations (14):
- Japan (14):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aichi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hokkaido
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyōgo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ibaraki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kyoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagano
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Okayama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saitama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toyama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wakayama

RESULTS

PARTICIPANT FLOW:
Groups:
- LY2189265 + Alpha-glucosidas e Inhibitor (a-GI): LY2189265: 0.75 mg administered SC, once weekly for 52 weeks
  Participants were to continue on their stable, pre-study, physician-prescribed dose of a-GI monotherapy throughout the study.
- LY2189265 + Thiazolidin Edione (TZD): LY2189265: 0.75 mg administered SC, once weekly for 52 weeks
  Participants were to continue on their stable, pre-study, physician-prescribed dose of TZD monotherapy throughout the study.
Period: Overall Study
Arm/Group | LY2189265 + Sulfonylureas (SU) | LY2189265 + Biguanides (BG) | LY2189265 + Alpha-glucosidas e Inhibitor (a-GI) | LY2189265 + Thiazolidin Edione (TZD) | LY2189265 + Glinides
Started | 131 | 61 | 65 | 66 | 71
Received at Least 1 Dose of Study Drug | 131 | 61 | 65 | 66 | 71
Completed | 121 | 59 | 57 | 63 | 66
Not Completed | 10 | 2 | 8 | 3 | 5
Not completed — Adverse Event | 8 | 1 | 6 | 2 | 2
Not completed — Protocol Violation | 2 | 0 | 1 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- LY2189265 + SU: LY2189265: 0.75 mg administered SC, once weekly for 52 weeks
  Participants were to continue on their stable, pre-study, physician-prescribed dose of SU monotherapy throughout the study.
- LY2189265 + BG: LY2189265: 0.75 mg administered SC, once weekly for 52 weeks
  Participants were to continue on their stable, pre-study, physician-prescribed dose of BG monotherapy throughout the study.
- LY2189265 + a-GI: LY2189265: 0.75 mg administered SC, once weekly for 52 weeks
  Participants were to continue on their stable, pre-study, physician-prescribed dose of a-GI monotherapy throughout the study.
- LY2189265 + TZD: LY2189265: 0.75 mg administered SC, once weekly for 52 weeks
  Participants were to continue on their stable, pre-study, physician-prescribed dose of TZD monotherapy throughout the study.
- Total: Total of all reporting groups
Arm/Group | LY2189265 + SU | LY2189265 + BG | LY2189265 + a-GI | LY2189265 + TZD | LY2189265 + Glinides | Total
Number analyzed (Participants) | 131 | 61 | 65 | 66 | 71 | 394
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.68 (11.59) | 52.69 (10.19) | 59.13 (10.51) | 56.40 (10.51) | 58.17 (10.30) | 57.35 (10.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 21 | 10 | 14 | 17 | 98
  Male | 95 | 40 | 55 | 52 | 54 | 296
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 131 | 61 | 65 | 66 | 71 | 394
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Japan | 131 | 61 | 65 | 66 | 71 | 394

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: A TEAE was defined as an event that first occurs or worsens (increases in severity) after baseline, regardless of causality or severity. The percentage of participants with TEAEs was calculated by dividing the number of participants with at least 1 TEAE over the 52-week treatment period by the total number of participants analyzed, multiplied by 100%. A summary of serious and other non-serious adverse events, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Baseline through 52 Weeks
Population: All enrolled participants who received at least 1 dose of study drug
Measure: Number; unit: percentage of participants
Arm/Group | LY2189265 + SU | LY2189265 + BG | LY2189265 + a-GI | LY2189265 + TZD | LY2189265 + Glinides
Number analyzed (Participants) | 131 | 61 | 65 | 66 | 71
percentage of participants | 85.5 | 83.6 | 70.8 | 80.3 | 73.2

2. Primary Outcome: Percentage of Participants With Hypoglycemic Episodes
Description: The percentage of participants with hypoglycemic episodes was calculated by dividing the number of participants with at least 1 hypoglycemic episode over the 52-week treatment period by the total number of participants analyzed, multiplied by 100%. All classifications of hypoglycemia (documented symptomatic, asymptomatic, severe, nocturnal, non-nocturnal, probable symptomatic, relative, and unspecified) were included, except for episodes of relative hypoglycemia that were not severe. A summary of serious and other non-serious adverse events, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Baseline through 52 Weeks
Population: All enrolled participants who received at least 1 dose of study drug
Measure: Number; unit: percentage of participants
Arm/Group | LY2189265 + SU | LY2189265 + BG | LY2189265 + a-GI | LY2189265 + TZD | LY2189265 + Glinides
Number analyzed (Participants) | 131 | 61 | 65 | 66 | 71
percentage of participants | 33.6 | 3.3 | 6.2 | 6.1 | 9.9

3. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c)
Time Frame: Baseline, up to 26 Weeks and up to 52 Weeks
Population: Participants who were randomized and received at least 1 dose of study drug with evaluable HbA1c data. Last observation carried forward (LOCF) was used to impute missing postbaseline values.
Measure: Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | LY2189265 + SU | LY2189265 + BG | LY2189265 + a-GI | LY2189265 + TZD | LY2189265 + Glinides
Number analyzed (Participants) | 131 | 61 | 65 | 66 | 71
percentage of HbA1c
  26 Weeks | -1.93 (0.09) | -1.58 (0.11) | -1.67 (0.10) | -1.71 (0.13) | -1.80 (0.12)
  52 Weeks | -1.67 (0.09) | -1.57 (0.11) | -1.65 (0.11) | -1.69 (0.13) | -1.65 (0.13)
Statistical Analysis 1: Comparison: LY2189265 + SU vs LY2189265 + BG vs LY2189265 + a-GI vs LY2189265 + TZD vs LY2189265 + Glinides; HbA1c at 26 Weeks; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; p-values are from within-group change t-test at the level of 0.05; Mean Difference (Final Values) = -1.77, 95% CI 2-sided [-1.87 to -1.67]
Statistical Analysis 2: Comparison: LY2189265 + SU vs LY2189265 + BG vs LY2189265 + a-GI vs LY2189265 + TZD vs LY2189265 + Glinides; HbA1c at 52 Weeks; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; p-values are from within-group change t-test at the level of 0.05; Mean Difference (Final Values) = -1.65, 95% CI 2-sided [-1.75 to -1.55]

4. Secondary Outcome: Percentage of Participants Who Achieve HbA1c ≤6.5% or <7%
Time Frame: 26 weeks and 52 weeks
Population: Participants who were randomized and received at least 1 dose of study drug with evaluable HbA1c data. LOCF was used to impute missing postbaseline values.
Measure: Number; unit: percentage of participants
Arm/Group | LY2189265 + SU | LY2189265 + BG | LY2189265 + a-GI | LY2189265 + TZD | LY2189265 + Glinides
Number analyzed (Participants) | 131 | 61 | 65 | 66 | 71
percentage of participants
  HbA1c ≤6.5% at Week 26 | 35.1 | 54.1 | 72.3 | 60.6 | 53.5
  HbA1c ≤6.5% at Week 52 | 31.3 | 57.4 | 70.8 | 57.6 | 47.9
  HbA1c <7.0% at Week 26 | 61.8 | 73.8 | 81.5 | 72.7 | 69.0
  HbA1c <7.0% at Week 52 | 48.9 | 73.8 | 83.1 | 77.3 | 62.0

5. Secondary Outcome: Change From Baseline in Fasting Blood Glucose (FBG)
Time Frame: Baseline, up to 26 weeks and up to 52 weeks
Population: Participants who were randomized and received at least 1 dose of study drug with evaluable FBG data. LOCF was used to impute missing postbaseline values.
Measure: Mean (Standard Error); unit: milligrams/deciliters (mg/dL)
Arm/Group | LY2189265 + SU | LY2189265 + BG | LY2189265 + a-GI | LY2189265 + TZD | LY2189265 + Glinides
Number analyzed (Participants) | 131 | 61 | 65 | 66 | 71
milligrams/deciliters (mg/dL)
  26 Weeks | -46.8 (4.2) | -37.9 (4.0) | -46.8 (4.7) | -42.1 (4.5) | -42.7 (3.9)
  52 Weeks | -43.2 (3.8) | -36.0 (4.2) | -47.0 (4.7) | -39.6 (5.0) | -45.8 (4.0)
Statistical Analysis 1: Comparison: LY2189265 + SU vs LY2189265 + BG vs LY2189265 + a-GI vs LY2189265 + TZD vs LY2189265 + Glinides; FBG at 26 Weeks; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; p-values are from within-group change t-test at the level of 0.05; Median Difference (Final Values) = -43.9, 95% CI 2-sided [-47.8 to -40.0]
Statistical Analysis 2: Comparison: LY2189265 + SU vs LY2189265 + BG vs LY2189265 + a-GI vs LY2189265 + TZD vs LY2189265 + Glinides; FBG at 52 Weeks; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; p-values are from within-group change t-test at the level of 0.05; Mean Difference (Final Values) = -42.6, 95% CI 2-sided [-46.4 to -38.7]

6. Secondary Outcome: Change From Baseline in 7-Point Self-Monitored Blood Glucose (SMBG)
Description: Participants were to test and record SMBG concentrations in their study diaries before each meal (breakfast, lunch, and dinner), approximately 2 hours after the start of each meal. For the mean of all 7-point blood glucose values, the daily mean was calculated as the average of 7 blood glucose values collected on a particular day. The mean of all 7-point blood glucose values at each visit was calculated as the average of 2 daily means. The change from baseline was calculated as the mean of all 7-point blood glucose values at endpoint minus the mean of all 7-point blood glucose values at baseline.
Time Frame: Baseline, up to 26 weeks and up to 52 weeks
Population: Participants who were randomized and received at least 1 dose of study drug with evaluable SMBG data. LOCF was used to impute missing postbaseline. values.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | LY2189265 + SU | LY2189265 + BG | LY2189265 + a-GI | LY2189265 + TZD | LY2189265 + Glinides
Number analyzed (Participants) | 131 | 61 | 65 | 66 | 71
mg/dL
  Pre-morning mean at 26 Weeks (n=131,61,64,66,71) | -44.70 (4.57) | -34.60 (3.88) | -45.97 (4.99) | -35.40 (3.85) | -48.26 (4.33)
  Pre-morning mean at 52 Weeks (n=131,61,64,66,71) | -42.93 (3.89) | -37.19 (3.83) | -45.69 (5.05) | -39.83 (4.24) | -46.45 (4.30)
  2hr postmorning meal at 26Weeks(n=131,61,65,66,71) | -69.66 (5.69) | -64.23 (6.35) | -73.43 (6.70) | -65.73 (5.94) | -67.99 (7.24)
  2hr postmorning meal at 52Weeks(n=131,61,65,66,71) | -58.50 (5.63) | -63.81 (7.22) | -73.62 (7.27) | -67.51 (6.49) | -73.78 (7.95)
  Pre-midday meal at 26 Weeks (n=131,61,65,66,71) | -49.95 (4.85) | -26.26 (4.93) | -54.75 (6.24) | -51.80 (6.68) | -54.51 (5.79)
  Pre-midday meal at 52 Weeks (n=131,61,65,66,71) | -43.90 (5.15) | -33.34 (5.12) | -55.96 (6.42) | -50.21 (7.04) | -56.07 (5.60)
  2hr postmidday meal at 26 Weeks(n=131,60,65,66,71) | -67.24 (5.24) | -50.03 (5.70) | -67.70 (7.37) | -80.02 (7.93) | -68.49 (7.84)
  2hr postmidday meal at 52 Weeks(n=131,60,65,66,71) | -57.27 (5.44) | -52.70 (5.26) | -63.47 (7.12) | -81.64 (8.68) | -65.46 (7.23)
  Pre-evening meal at 26 Weeks (n=130,61,65,66,70) | -44.57 (5.63) | -25.66 (5.28) | -57.82 (6.83) | -43.22 (7.53) | -46.85 (5.88)
  Pre-evening meal at 52 Weeks (n=130,61,65,66,70) | -43.90 (5.39) | -25.34 (5.55) | -54.66 (7.35) | -42.15 (7.44) | -51.64 (6.10)
  2hr postevening meal at 26Weeks(n=128,61,65,66,69) | -62.24 (6.05) | -45.41 (6.71) | -71.15 (7.57) | -66.14 (8.22) | -68.75 (7.88)
  2hr postevening meal at 52Weeks(n=128,61,65,66,69) | -58.98 (5.71) | -48.61 (6.45) | -63.82 (7.00) | -69.30 (8.60) | -64.22 (7.07)
  Bedtime at 26 Weeks (n=128, 61, 65, 63, 67) | -61.07 (5.08) | -49.98 (6.48) | -63.98 (6.90) | -66.19 (8.75) | -64.01 (6.56)
  Bedtime at 52 Weeks (n=128, 61, 65, 63, 67) | -54.07 (5.24) | -52.70 (6.45) | -66.74 (7.31) | -68.42 (9.05) | -64.41 (6.21)
Statistical Analysis 1: Comparison: LY2189265 + SU vs LY2189265 + BG vs LY2189265 + a-GI vs LY2189265 + TZD vs LY2189265 + Glinides; Pre-morning meal at 26 Weeks; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; p-values are from within-group change t-test at the level of 0.05; Mean Difference (Final Values) = -42.42, 95% CI 2-sided [-46.55 to -38.29]
Statistical Analysis 2: Comparison: LY2189265 + SU vs LY2189265 + BG vs LY2189265 + a-GI vs LY2189265 + TZD vs LY2189265 + Glinides; Pre-morning meal at 52 Weeks; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; p-values are from within-group change t-test at the level of 0.05; Mean Difference (Final Values) = -42.60, 95% CI 2-sided [-46.44 to -38.76]
Statistical Analysis 3: Comparison: LY2189265 + SU vs LY2189265 + BG vs LY2189265 + a-GI vs LY2189265 + TZD vs LY2189265 + Glinides; 2 hours post-morning meal at 26 Weeks; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; p-values are from within-group change t-test at the level of 0.05; Mean Difference (Final Values) = -68.48, 95% CI 2-sided [-74.18 to -62.79]
Statistical Analysis 4: Comparison: LY2189265 + SU vs LY2189265 + BG vs LY2189265 + a-GI vs LY2189265 + TZD vs LY2189265 + Glinides; 2 hours post-morning meal at 52 Weeks; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; p-values are from within-group change t-test at the level of 0.05; Mean Difference (Final Values) = -66.08, 95% CI 2-sided [-72.12 to -60.04]
Statistical Analysis 5: Comparison: LY2189265 + SU vs LY2189265 + BG vs LY2189265 + a-GI vs LY2189265 + TZD vs LY2189265 + Glinides; Pre-midday meal at 26 Weeks; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; p-values are from within-group change t-test at the level of 0.05; Mean Difference (Final Values) = -48.21, 95% CI 2-sided [-53.32 to -43.09]
Statistical Analysis 6: Comparison: LY2189265 + SU vs LY2189265 + BG vs LY2189265 + a-GI vs LY2189265 + TZD vs LY2189265 + Glinides; Pre-midday meal at 52 Weeks; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; p-values are from within-group change t-test at the level of 0.05; Mean Difference (Final Values) = -47.51, 95% CI 2-sided [-52.77 to -42.24]
Statistical Analysis 7: Comparison: LY2189265 + SU vs LY2189265 + BG vs LY2189265 + a-GI vs LY2189265 + TZD vs LY2189265 + Glinides; 2 hours post-midday meal at 26 Weeks; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; p-values are from within-group change t-test at the level of 0.05; Mean Difference (Final Values) = -67.06, 95% CI 2-sided [-73.02 to -61.11]
Statistical Analysis 8: Comparison: LY2189265 + SU vs LY2189265 + BG vs LY2189265 + a-GI vs LY2189265 + TZD vs LY2189265 + Glinides; 2 hours post-midday meal at 52 Weeks; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; p-values are from within-group change t-test at the level of 0.05; Mean Difference (Final Values) = -63.17, 95% CI 2-sided [-69.16 to -57.18]
Statistical Analysis 9: Comparison: LY2189265 + SU vs LY2189265 + BG vs LY2189265 + a-GI vs LY2189265 + TZD vs LY2189265 + Glinides; Pre-evening meal at 26 Weeks; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; p-values are from within-group change t-test at the level of 0.05; Mean Difference (Final Values) = -44.00, 95% CI 2-sided [-49.67 to -38.34]
Statistical Analysis 10: Comparison: LY2189265 + SU vs LY2189265 + BG vs LY2189265 + a-GI vs LY2189265 + TZD vs LY2189265 + Glinides; Pre-evening meal at 52 Weeks; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; p-values are from within-group change t-test at the level of 0.05; Mean Difference (Final Values) = -43.88, 95% CI 2-sided [-49.55 to -38.21]
Statistical Analysis 11: Comparison: LY2189265 + SU vs LY2189265 + BG vs LY2189265 + a-GI vs LY2189265 + TZD vs LY2189265 + Glinides; 2 hours post-evening meal at 26 Weeks; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; p-values are from within-group change t-test at the level of 0.05; Mean Difference (Final Values) = -62.91, 95% CI 2-sided [-69.32 to -56.50]
Statistical Analysis 12: Comparison: LY2189265 + SU vs LY2189265 + BG vs LY2189265 + a-GI vs LY2189265 + TZD vs LY2189265 + Glinides; 2 hours post-evening meal at 52 Weeks; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; p-values are from within-group change t-test at the level of 0.05; Mean Difference (Final Values) = -60.84, 95% CI 2-sided [-66.95 to -54.74]
Statistical Analysis 13: Comparison: LY2189265 + SU vs LY2189265 + BG vs LY2189265 + a-GI vs LY2189265 + TZD vs LY2189265 + Glinides; Bedtime meal at 26 Weeks; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; p-values are from within-group change t-test at the level of 0.05; Mean Difference (Final Values) = -61.15, 95% CI 2-sided [-66.93 to -55.37]
Statistical Analysis 14: Comparison: LY2189265 + SU vs LY2189265 + BG vs LY2189265 + a-GI vs LY2189265 + TZD vs LY2189265 + Glinides; Bedtime meal at 52 Weeks; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; p-values are from within-group change t-test at the level of 0.05; Mean Difference (Final Values) = -60.16, 95% CI 2-sided [-66.07 to -54.25]

7. Secondary Outcome: Change From Baseline in Body Weight
Time Frame: Baseline, up to 26 weeks and up to 52 weeks
Population: Participants who were randomized and received at least 1 dose of study drug with evaluable body weight data. LOCF was used to impute missing postbaseline values.
Measure: Mean (Standard Error); unit: kilograms (kg)
Arm/Group | LY2189265 + SU | LY2189265 + BG | LY2189265 + a-GI | LY2189265 + TZD | LY2189265 + Glinides
Number analyzed (Participants) | 131 | 61 | 65 | 66 | 71
kilograms (kg)
  26 Weeks | 0.02 (0.22) | -0.74 (0.39) | -1.22 (0.33) | 0.78 (0.30) | 0.19 (0.25)
  52 Weeks | 0.10 (0.24) | -0.87 (0.40) | -1.24 (0.42) | 1.02 (0.35) | 0.04 (0.26)
Statistical Analysis 1: Comparison: LY2189265 + SU vs LY2189265 + BG vs LY2189265 + a-GI vs LY2189265 + TZD vs LY2189265 + Glinides; Body weight at 26 Weeks; Test type: Superiority or Other; p < 0.277, t-test, 2 sided; p-values are from within-group change t-test at the level of 0.05; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-0.40 to 0.12]
Statistical Analysis 2: Comparison: LY2189265 + SU vs LY2189265 + BG vs LY2189265 + a-GI vs LY2189265 + TZD vs LY2189265 + Glinides; Body weight at 52 Weeks; Test type: Superiority or Other; p = 0.382, t-test, 2 sided; p-values are from within-group change t-test at the level of 0.05; Mean Difference (Final Values) = -0.13, 95% CI 2-sided [-0.42 to 0.16]

8. Secondary Outcome: Change From Baseline in Updated Homeostasis Model Assessment (HOMA2)
Description: The HOMA2 is a computer model that uses fasting plasma insulin and glucose concentrations to estimate steady state pancreatic beta cell function (%B) and to estimate insulin sensitivity (%S) as a percentage of a normal reference population (normal young adults). The normal reference population was set at 100%. The change from baseline for fasting insulin concentrations are presented as insulin secretion (HOMA2-%B) and insulin sensitivity (HOMA2-%S).
Time Frame: Baseline, up to 26 weeks and up to 52 weeks
Population: Participants who were randomized and received at least 1 dose of study drug with evaluable HOMA2 data. LOCF was used to impute missing postbaseline values.
Measure: Mean (Standard Error); unit: percentage of HOMA2
Arm/Group | LY2189265 + SU | LY2189265 + BG | LY2189265 + a-GI | LY2189265 + TZD | LY2189265 + Glinides
Number analyzed (Participants) | 127 | 59 | 62 | 59 | 64
percentage of HOMA2
  HOMA2-%B, 26 Weeks | 29.10 (2.75) | 28.15 (2.79) | 30.88 (3.25) | 27.34 (2.60) | 26.93 (2.59)
  HOMA2-%B, 52 Weeks | 26.06 (2.77) | 26.05 (2.97) | 28.06 (3.61) | 25.38 (2.53) | 33.51 (3.81)
  HOMA2-%S, 26 Weeks | -4.80 (3.40) | -3.48 (4.39) | 7.57 (5.60) | -5.50 (5.21) | -4.41 (4.05)
  HOMA2-%S, 52 Weeks | -3.99 (3.18) | -3.83 (4.89) | 6.86 (5.24) | 0.47 (5.87) | -5.51 (4.71)
Statistical Analysis 1: Comparison: LY2189265 + SU vs LY2189265 + BG vs LY2189265 + a-GI vs LY2189265 + TZD vs LY2189265 + Glinides; HOMA2-B% at 26 Weeks; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; p-values are from within-group change t-test at the level of 0.05; Mean Difference (Final Values) = 28.59, 95% CI 2-sided [26.00 to 31.18]
Statistical Analysis 2: Comparison: LY2189265 + SU vs LY2189265 + BG vs LY2189265 + a-GI vs LY2189265 + TZD vs LY2189265 + Glinides; HOMA2-B% at 52 Weeks; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; p-values are from within-group change t-test at the level of 0.05; Mean Difference (Final Values) = 27.57, 95% CI 2-sided [24.73 to 30.41]
Statistical Analysis 3: Comparison: LY2189265 + SU vs LY2189265 + BG vs LY2189265 + a-GI vs LY2189265 + TZD vs LY2189265 + Glinides; HOMA2-S% at 26 Weeks; Test type: Superiority or Other; p = 0.194, t-test, 2 sided; p-values are from within-group change t-test at the level of 0.05; Mean Difference (Final Values) = -2.57, 95% CI 2-sided [-6.46 to 1.32]
Statistical Analysis 4: Comparison: LY2189265 + SU vs LY2189265 + BG vs LY2189265 + a-GI vs LY2189265 + TZD vs LY2189265 + Glinides; HOMA2-S% at 52 Weeks; Test type: Superiority or Other; p = 0.400, t-test, 2 sided; p-values are from within-group change t-test at the level of 0.05; Mean Difference (Final Values) = -1.70, 65% CI 2-sided [-5.68 to 2.27]

ADVERSE EVENTS:
Arm/Group | LY2189265 + SU | LY2189265 + BG | LY2189265 + a-GI | LY2189265 + TZD | LY2189265 + Glinides
Serious Adverse Events (participants affected / at risk) | 9/131 | 3/61 | 4/65 | 1/66 | 3/71
Other Adverse Events (participants affected / at risk) | 112/131 | 51/61 | 46/65 | 53/66 | 52/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | LY2189265 + SU (N=131) | LY2189265 + BG (N=61) | LY2189265 + a-GI (N=65) | LY2189265 + TZD (N=66) | LY2189265 + Glinides (N=71)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pancreatic enzyme abnormality (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign soft tissue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/36 (0) | 0/21 (0) | 1/10 (1) | 0/14 (0) | 0/17 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 0/95 (0) | 1/40 (1) | 0/55 (0) | 0/52 (0) | 0/54 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | LY2189265 + SU (N=131) | LY2189265 + BG (N=61) | LY2189265 + a-GI (N=65) | LY2189265 + TZD (N=66) | LY2189265 + Glinides (N=71)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Polycythaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Tachycardia (Cardiac disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deafness neurosensory (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear pruritus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Basedow's disease (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blepharitis (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic retinopathy (Eye disorders) | 4 (4) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Dry eye (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Iritis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Macular oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Optic ischaemic neuropathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 2 (4) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 4 (8) | 0 (0) | 2 (2) | 2 (2) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Abdominal tenderness (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute abdomen (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 20 (22) | 3 (3) | 8 (8) | 3 (3) | 5 (6)
Dental caries (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 13 (14) | 9 (13) | 3 (3) | 5 (8) | 7 (9)
Dyspepsia (Gastrointestinal disorders) | 6 (18) | 2 (2) | 1 (2) | 0 (0) | 5 (8)
Eructation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Faeces hard (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 4 (4) | 3 (3) | 2 (2) | 3 (3) | 2 (2)
Gastritis atrophic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal hypomotility (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3) | 1 (1) | 3 (4) | 1 (1) | 2 (2)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 17 (82) | 2 (2) | 4 (8) | 5 (6) | 3 (3)
Pancreatic enzyme abnormality (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 8 (11) | 1 (1) | 3 (3) | 3 (5) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Facial pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Feeling abnormal (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site eczema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Injection site haemorrhage (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site induration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Injection site pruritus (General disorders) | 2 (4) | 0 (0) | 2 (2) | 3 (3) | 3 (3)
Injection site reaction (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Local swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Xerosis (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gallbladder polyp (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hepatic cyst (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Hepatitis alcoholic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Adenoiditis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 10 (14) | 1 (1) | 0 (0) | 2 (4) | 2 (2)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic sinusitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Eczema infected (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enteritis infectious (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 2 (4) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Genital herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Helicobacter infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 6 (6) | 7 (7) | 0 (0) | 0 (0) | 3 (3)
Nasopharyngitis (Infections and infestations) | 31 (51) | 16 (25) | 11 (15) | 16 (26) | 16 (18)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periodontitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 7 (8) | 2 (2) | 3 (3) | 6 (6) | 0 (0)
Pulpitis dental (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 4 (4) | 1 (1) | 2 (2) | 2 (2)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heat stroke (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 3 (4) | 0 (0) | 2 (2) | 2 (2) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Blood pressure decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure diastolic increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood uric acid increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 11 (11) | 6 (6) | 6 (7) | 3 (3) | 2 (2)
Pancreatic enzymes increased (Investigations) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 10 (16) | 3 (3) | 3 (3) | 1 (1) | 2 (2)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 2 (2) | 2 (2) | 6 (7) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Knee deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nodal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Soft tissue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carotid arteriosclerosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 4 (5) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lacunar infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 2 (17) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Trigeminal neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Visual field defect (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased interest (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cystitis haemorrhagic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic nephropathy (Renal and urinary disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amenorrhoea (Reproductive system and breast disorders) | 0/36 (0) | 1/21 (1) | 0/10 (0) | 0/14 (0) | 0/17 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 1/95 (1) | 0/40 (0) | 0/55 (0) | 0/52 (0) | 0/54 (0)
Prostatitis (Reproductive system and breast disorders) | 1/95 (1) | 0/40 (0) | 0/55 (0) | 0/52 (0) | 0/54 (0)
Pruritus genital (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Varicocele (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cold urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (1) | 2 (2) | 0 (0) | 2 (3)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukoplakia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Onychalgia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palmoplantar keratoderma (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Perivascular dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (6) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Xeroderma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder catheterisation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon polypectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary angioplasty (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery bypass (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dental care (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal sphincterotomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Open reduction of fracture (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Percutaneous coronary intervention (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Photocoagulation (Surgical and medical procedures) | 1 (3) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Skin lesion excision (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 5 (5) | 3 (3) | 4 (4) | 2 (2) | 3 (3)
Peripheral coldness (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days